CLINICAL TRIAL: NCT06070922
Title: Role Of LDCT Chest In Assessment Of Apparently Healthy Smokers
Brief Title: LDCT Chest In Assessment Of Apparently Healthy Smokers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Lecture of chest diseases, Assiut University
Other Study IDs: Low Dose CT & healthy smoker
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effectiveness of LDCT screening in detecting early-stage lung cancers among smokers who do not have symptoms of lung disease.

DETAILED DESCRIPTION:
Tobacco smoking is the leading preventable cause of death worldwide .Chronic Obstructive Pulmonary Disease (COPD), lung cancer, and cardiovascular disease will be responsible for the majority of deaths in the developed world in the coming decades .

COPD is characterised by chronic airflow limitation caused by a combination of small airway inflammation and parenchymal destruction (emphysema) . Since computed tomography (CT) has been validated as a non-invasive technique capable of identifying areas of lung parenchyma with emphysema , several studies have identified a subgroup of apparently healthy smokers who have emphysema but no airway obstruction Furthermore, this subgroup has the highest risk of developing lung cancer among smokers .It has been proposed that systemic inflammation may play an important pathogenic role in carcinogenesis . We will conducted this cross sectional study between. current and former smokers without airway obstruction participating in a lung cancer screening study: a study group of smokers with emphysema on the CT, and a control group of smokers without emphysema.

ELIGIBILITY:
Inclusion Criteria:

- Participants have at least 45years old had smoked 10 pack-years or more

Exclusion Criteria:

* Age: less than 45 years. Non smoker Evidence of airway obstruction by Pulmonery Function Test

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After taking the informed consent, full history will be taken from all patients participating in the study include smoking history. Detailed clinical examination and routine laboratory investigations will be done.
  Low Dose CT chest( reduced the radiation exposure to 1.6 mSv ) will be done . Spirometry spirometry will be performed using standard techniques according to ATS-ERS criteria 2019 .
  These individuals will further classified into two groups according to the presence or absence of emphysema on the LDCT, the study group have smokers and former smokers with emphysema on the LDCT but no evidence of airway obstruction, whereas the comparison group current and former smokers without emphysema and without obstruction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
• Prevalence of Emphysema in apparently healthy smoker • Association between lung cancer and emphysema • Rate of early-stage lung cancer detection (Stage I/II) • Lung cancer mortality rate | baseline
  from LDCT Chest

SECONDARY OUTCOMES:
Diagnostic accuracy and performance of LDCT • Positive predictive value of LDCT screening • Rate of incidental findings on LDCT requiring follow up • Rate of unnecessary invasive procedures due to false positives | baseline
  by Statistical tests and anylasis

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa sayed, lecture, Study Chair — Assiut University

REFERENCES:
- [Background] Koyama H, Ohno Y, Yamazaki Y, Matsumoto K, Onishi Y, Takenaka D, Yoshikawa T, Nishio M, Matsumoto S, Murase K, Nishimura Y, Sugimura K. Reduced-dose chest CT with 3D automatic exposure control vs. standard chest CT: quantitative assessment of emphysematous changes in smokers' lung parenchyma. Eur J Radiol. 2012 Jun;81(6):1330-4. doi: 10.1016/j.ejrad.2011.03.037. Epub 2011 Jun 24. PMID 21703788
- [Background] Bonney A, Malouf R, Marchal C, Manners D, Fong KM, Marshall HM, Irving LB, Manser R. Impact of low-dose computed tomography (LDCT) screening on lung cancer-related mortality. Cochrane Database Syst Rev. 2022 Aug 3;8(8):CD013829. doi: 10.1002/14651858.CD013829.pub2. PMID 35921047